CLINICAL TRIAL: NCT04440072
Title: Comparison of 3 Ultrasonic Techniques for Measuring the Systolic Pressure Index
Acronym: ABIPULSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 20-037
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Peripheral Arterial Disease; Atherosclerosis Obliterans; Atherosclerosis Right Leg; Atherosclerosis Left Leg
Keywords: ankle brachial index; color duplex ultrasound; pulsed doppler
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Continuous Doppler ankle brachial index (ABI) is the gold standard for screening and monitoring of peripheral arterial disease (PAD) but is no longer carried out in clinical practice.

The recommended measurement was gradually replaced by colour or pulsed Doppler without validation of these techniques.

The objective of our study is to compare these two techniques (color Doppler and pulsed Doppler in echodoppler) with respect to the gold standard (continuous Doppler) for ABI measurement.

ELIGIBILITY:
Inclusion Criteria:

Patient referred to the Vascular Medicine Department of Caen University Hospital for a vascular examination with ABI measurement having been informed and not objecting to participation in the study and benefiting from a social protection system.

Exclusion Criteria:

* Patient with arrhythmia
* Patient with trans-tibial or more proximal amputation
* Patient with extensive trophic disorder not allowing measurement
* Patient with subgonal bypass
* Known bilateral sub-clavian stenoses
* Patient deprived of liberty or under a measure of legal protection
* Interned patient for the treatment of a psychiatric or physical illness
* Patients who are legally incompetent, under the protection of justice, under guardianship or trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient referred to the Vascular Medicine Department for a vascular examination with ABI measurement. In most cases, these patients present with symptoms suggestive of PAD, most often with vascular risk factors for atherosclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-06-22 (Estimated); Study Completion 2021-06-22 (Estimated)

PRIMARY OUTCOMES:
Concordance on the IPS value measured with pulsed Doppler compared to gold standard | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided